CLINICAL TRIAL: NCT07255209
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Clinical Trial to Assess the Efficacy and Safety of IBI362 in Chinese Adolescents With Obesity or Overweight（GLORY-YOUNG）
Brief Title: A Study of IBI362 in Chinese Adolescents With Obesity or Overweight
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362B304
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Adolescents With Obesity or Overweight With Weight-Related Comorbidities
MeSH Terms: interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- IBI362-dose2 (Experimental)
  Interventions: Drug: IBI362
- IBI362-dose1 (Experimental)
  Interventions: Drug: IBI362

INTERVENTIONS:
Drug: Placebo — Placebo SA.QW
  Arms: Placebo
Drug: IBI362 — IBI362 SA.QW
  Arms: IBI362-dose1; IBI362-dose2

SUMMARY:
The study is designed to assess the efficacy and safety of multiple doses of IBI362 in Chinese adolescent subjects with obesity or overweight. It plans to enroll 180 adolescents (aged ≥12 and <18 years) who have failed to achieve a 5 kg weight reduction after at least 12 weeks of dietary and exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be enrolled:

Key Inclusion Criteria：

1. Male or female participants aged ≥12 years and <18 years at the time of signing the informed consent/assent form.
2. BMI at screening meeting the obesity criteria defined by "WS/T 586-2018 Screening for Overweight and Obesity in School-Age Children and Adolescents" or meeting overweight criteria plus at least one weight-related comorbidity: prediabetes, type 2 diabetes, hypertension, dyslipidemia, fatty liver disease, or obstructive sleep apnea syndrome.
3. Weight change <5 kg after ≥12 weeks of diet and exercise alone before screening (per self/parental report).

Exclusion Criteria:

Key Exclusion Criteria：

1. Prior diagnosis of type 1 diabetes.
2. Pre-pubertal participants (Tanner Stage I).
3. History of (or planned) bariatric surgery (except liposuction/abdominoplasty or acupuncture for weight loss performed >1 year before screening).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in BMI | Week 32

SECONDARY OUTCOMES:
Percentage of Participants with ≥5% BMI Reduction | Week 32
Percent Change from Baseline in BMI | Week 52
Percentage of Participants with ≥5% BMI Reduction | Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China